CLINICAL TRIAL: NCT02700490
Title: Evaluating the Clinical Cost-effectiveness of Two Primary Mental Health Service Frameworks in Yogyakarta, Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Universita di Verona (Other); Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Sabrina Anjara, PhD, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRE.2015.108
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy

ARMS (2):
- Specialist (Active Comparator): Assessment and treatment of common mental disorders by a clinical psychologist in primary care facilities.
  Interventions: Behavioral: Psychotherapy
- Enhanced Usual Care (Experimental): Assessment and treatment of common mental disorders by a general practitioner and nurse practitioner, who have been trained in the WHO mhGap manual, in primary care facilities.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Behaviour Therapy or Cognitive Behaviour Therapy which forms "service as usual" in primary care centres in Indonesia.

SUMMARY:
This study is a cluster randomised controlled trial, which aims to examine the short-term strategy of addressing treatment gap through increasing primary mental health service capacity. This study aims to compare after 6 months and 12 months, the effectiveness of a specialist model of mental health care and an enhanced usual care (task-sharing) framework, in terms of reducing mental health symptoms, reducing disability, and improving quality of life, as well as the health services costs (and potentially societal costs) associated with these outcomes in 400 patients.

DETAILED DESCRIPTION:
Two primary mental health service frameworks in Yogyakarta are compared: the specialist framework and the enhanced usual care framework. Both frameworks have not been evaluated in the Indonesian context, despite their potential to be the framework of choice for other provincial and district governments to adopt. Extension to existing services has been planned, which provides us with the opportunity to implement in a random manner the enhanced usual care framework in new areas.

This study aims to compare after 6 months and 12 months, the effectiveness of a specialist model of mental health care and an enhanced usual care (task-sharing) framework, in terms of reducing mental health symptoms, reducing disability, and improving quality of life, as well as the health services costs (and potentially societal costs) associated with these outcomes in 400 patients. This study receives ground-level support from the Centre for Public Mental Health, Universitas Gadjah Mada, which manages the specialist primary mental health framework in Yogyakarta province, regional and national-level support from the Ministry of Health of Indonesia, and will be hopefully funded by the LPDP, Ministry of Finance of Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Participants are adults who meet the screening criteria for depression and anxiety on the self-report General Health Questionnaire (GHQ-12)

Exclusion Criteria:

* Potential participants who are currently receiving treatment for any mental health disorders will not be invited to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Health of Nations Outcomes Scale (HoNOS) score from baseline | Baseline, 6 months and 12 months
  Measures health and social functioning of participants
Change in Clinical Interview Schedule Revised (CIS-R) score from baseline | Baseline, 6 months and 12 months
  Measures the presence and severity of psychiatric symptoms

SECONDARY OUTCOMES:
Change in WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) score from baseline | Baseline, 6 months and 12 months
  Measures type and extent of disability of participants
Change in European Quality of Life Scale (EQ-5D) score from baseline | Baseline, 6 months and 12 months
  Measures quality of life of participants
Utility of service as measured by Client Service Receipt Inventory (CSRI) | Baseline, 6 months and 12 months
  Measures service utility within the time frame

CONTACTS AND LOCATIONS:
Overall Officials: Tine Van Bortel, Study Director — University of Cambridge; Carol Brayne, Study Chair — University of Cambridge
Locations (1):
- Centre for Public Mental Health, Yogyakarta, D.I Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the University of Cambridge data repository.
Supporting Information: Study Protocol
URL: https://www.protocols.io/view/evaluating-the-clinical-cost-effectiveness-of-two-6ythfwn

REFERENCES:
- [Derived] Anjara SG, Bonetto C, Ganguli P, Setiyawati D, Mahendradhata Y, Yoga BH, Trisnantoro L, Brayne C, Van Bortel T. Can General Practitioners manage mental disorders in primary care? A partially randomised, pragmatic, cluster trial. PLoS One. 2019 Nov 7;14(11):e0224724. doi: 10.1371/journal.pone.0224724. eCollection 2019. PMID 31697724
- Available data/document: Complete Data Set: 10.17863/CAM.43399 — https://doi.org/10.17863/CAM.43399